CLINICAL TRIAL: NCT03591783
Title: Impact of Sustained Virologic Response on Glycemic Control Among Diabetic Patients With Hepatitis C Virus Related Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Judy, Principal investigator, Assiut University
Other Study IDs: HCVDM
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis c
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: All patients will be subjected to: Baseline investigations, end of treatment investigations and 3 months after treatment investigations.

SUMMARY:
Hepatitis C virus (HCV) is a major cause of chronic liver disease. The World Health Organization has reported that 170 million people are chronically infected with HCV globally. The highest prevalence of HCV infection worldwide exists in Egypt (15%); 90% of infection among Egyptian patients is due to genotype 4

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection will be diagnosed based on positive testing for serum HCV RNA and anti-HCV Ab.
* Diagnosis of type 2 DM will depend on fasting level of serum glucose more than 126 mg/dl and/or serum level of HbA1c more than 6.5 % on oral hypoglycemic therapy.

Exclusion Criteria:

* Chronic hepatitis due to causes other than HCV infection
* Coinfection with HBV infection
* Hepatocellular carcinoma
* Child C stage of liver cirrhosis.
* Patients with type I diabetes mellitus.
* Cardiopulmonary diseases.
* Major illness.
* Patient receiving corticosteroids.
* Patient refused consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with chronic HCV infection with type 2 DM, who are eligible for antiviral therapy.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients with glycemic control | 3 months
  Exploring the impact of achieving SVR by directly acting antiviral drugs on glycemic control among diabetic patients with HCV infection.